CLINICAL TRIAL: NCT02945995
Title: Outcome After Arthroscopic Labrum Surgery in Patients Treated With Periacetabular Osteotomy
Brief Title: Outcome After Arthroscopic Surgery in Patients Treated With PAO
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, Aarhus University Hospital
Other Study IDs: CHA-PostPAO
Record Dates: First submitted 2015-03-18; First posted 2016-10-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-10

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: hip arthroscopy — Follow up after hip arthroscopy in pt with previous PAO. Follow up by questionnaires send til the cohort

SUMMARY:
The purpose of the study is to evaluate outcome after arthroscopy if the hip in patients previous treated with periacetabular osteotomy

DETAILED DESCRIPTION:
It is well known the patients with developmental dysplasia of the hip beyond the bony malformation has intraarticular damage to labrum and chondral structures.

In DK, if the patients has persistent pain in the hip joint after PAO, they have been offered a hip arthroscopy, however we do not if their hip functions and pain improved by the surgery

The investigator aimed to make a short to middle-term followup study to see if the patients had benefits of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* previous PAO and hip arthroscopy
* developmental dysplasia of the hip

Exclusion Criteria:

* calve legg perthes disease
* femoral osteotomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing hip arthrocopy previous treated with periacetabular osteotomy
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of patient with the need of a total hip arthroplasty after PAO and hip arthroscopy | 48 months after hip arthroscopy
  Questionnaire

SECONDARY OUTCOMES:
Evaluation of the patients pain in rest and during activity on a NRS Scale | 48 months after hip arthroscopy
  Questionnaire
Evaluation of hip function and pain using MHHS (modified harris hip score) | 48 months after hip arthroscopy
  Questionnaire
Evaluation of hip function and pain using HOS (Hip outcome score) | 48 months after hip arthroscopy
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lind, MD,PhD,DmSc, Study Director — Aarhus University Hospital